CLINICAL TRIAL: NCT00005071
Title: A Pilot Study Leading to a Randomized Trial Comparing Outcomes in Patients With Suspected Lung Cancer Investigated in the Conventional Locally (LO) Based (BA) Chest Clinic Compared With a Centralized 2 Stop Pathway (LOBA 2STOP)
Brief Title: Diagnosis and Treatment Planning in Patients Suspected of Having Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Diagnostic
Other Study IDs: CDR0000067676; RMNHS-PATHWAY; EU-99039
Record Dates: First submitted 2000-04-06; First posted 2004-04-19 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-06

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Biopsy; Bronchoscopy

INTERVENTIONS:
Procedure: biopsy
Procedure: bronchoscopy
Procedure: computed tomography
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Diagnostic procedures and treatment-planning systems may affect outcome in patients suspected of having lung cancer.

PURPOSE: Randomized diagnostic trial to compare the effectiveness of two types of diagnostic and treatment-planning systems in patients who are suspected of having lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the survival rate of patients with suspected lung cancer when diagnosed and managed using the conventional locally based approach versus a new centralized system using a 2 stop diagnosis. II. Compare the resection rate in both diagnostic arms. III. Assess the quality of service given in both diagnostic arms.

OUTLINE: This is a randomized study. Patients present to a general practitioner where they are referred to the local chest clinic. Patients are seen by the chest physician and, if deemed eligible, are randomized between 2 diagnostic arms. Arm I (Conventional Locally Based Diagnosis): Patients undergo bronchoscopy and CT scan as appropriate, and then are discussed or referred by individual chest physicians, as is the current practice. The optimal period for diagnosis and discussion of management plans is 6 weeks. Arm II (Centralized 2 Stop Diagnosis): Patients undergo CT scan the following Monday morning. The consultant radiologist advises the most appropriate diagnostic test (e.g., bronchoscopy or percutaneous needle biopsy) to be done that same Monday. A tissue diagnosis is available Thursday morning for the multidisciplinary meeting attended by the chest physician, medical and clinical oncologists, and a surgeon, and the patient treatment plan is decided. Quality of life is assessed at baseline and at 6 weeks. Patients are followed for 2 years.

PROJECTED ACCRUAL: A total of 252-315 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Possible diagnosis of lung cancer Fit enough for bronchoscopy and CT scan

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-10

CONTACTS AND LOCATIONS:
Overall Officials: Mary O'Brien, MD, Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, Sutton, England, United Kingdom